CLINICAL TRIAL: NCT05842291
Title: Personalized Brain Functional Sectors (pBFS) Guided High-dose rTMS Therapy for Treatment-resistant Depression: A Randomized, Double-Blind, Sham-controlled Trial
Brief Title: pBFS Guided High-dose rTMS Therapy for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLMDDhlg2
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Treatment-Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active rTMS with short inter-session interval (Experimental): Patients in this group will receive rTMS intervention with short inter-session intervals.
  Interventions: Device: Active rTMS with short inter-session interval
- Sham rTMS with short inter-session interval (Sham Comparator): Patients in this group will receive sham rTMS intervention with short inter-session intervals.
  Interventions: Device: Sham rTMS with short inter-session interval
- Active rTMS with long inter-session interval (Active Comparator): Patients in this group will receive rTMS intervention with long inter-session intervals.
  Interventions: Device: Active rTMS with long inter-session interval

INTERVENTIONS:
Device: Active rTMS with short inter-session interval — Participants in this group will receive ten sessions per day of 1800 pulses per session, at an inter-session interval of 20 min for 5 days. The individualized target will be generated using the personalized Brain Functional Sectors (pBFS) method.
  Arms: Active rTMS with short inter-session interval
Device: Sham rTMS with short inter-session interval — Participants in this group will receive ten sessions per day of 1800 pulses per session, at an inter-session interval of 20 min for 5 days, using sham stimulation coils that comprehensively mimic the active condition. The individualized target will be generated using the personalized Brain Functional Sectors (pBFS) method.
  Arms: Sham rTMS with short inter-session interval
Device: Active rTMS with long inter-session interval — Participants in this group will receive ten sessions per day of 1800 pulses per session, at an inter-session interval of 50 min for 5 days. The individualized target will be generated using the personalized Brain Functional Sectors (pBFS) method.
  Arms: Active rTMS with long inter-session interval

SUMMARY:
We aim to evaluate the safety and efficacy of pBFS-guided high-dose rTMS therapy with short inter-session interval for patients with treatment-resistant depression

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. Currently, the FDA cleared the SAINT Neuromodulation System for the treatment of Treatment-Resistant Depression(TRD) over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been effective in a short period of time for treatment-resistant depression. The limitation of this approach includes the long inter-session interval (~50min) of the treatment, patients need to wait about 8 hours for 10 session's intervention per day. Therefore, it is urgent to explore the efficacy and safety of rTMS with a short inter-session interval (e.g. 20 min) that is more acceptable for TRD patients.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 1:1:1 ratio to the active short-interval rTMS group, active short-interval rTMS group, and active long-interval rTMS group. Then all participants will undergo a 5 day rTMS modulation followed by a four-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized/outpatient patients aged 18-65 years (inclusive), male or female.
* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for the depression disorder without psychotic symptoms, and currently experiencing the first episode or recurrence episode.
* Total HAMD17 score ≥18 before randomization.
* Total MADRS score ≥20 before randomization.
* A stable or no-drug use for at least 4 weeks before randomization. The type and dose of the antidepressant regimen remained unchanged throughout the study.
* No response (symptom improvement≥50%) in previous treatments with at least two antidepressants for a full dose and full course.
* Voluntarily participate in the trial and sign informed consent. Able to comply with the planned visit, examination and treatment plan, and other study procedures.

Exclusion Criteria:

* Meet DSM-5 diagnostic criteria for other mental disorders (e.g., schizophrenia spectrum disorders, bipolar and related disorders, anxiety disorders, compulsion, and related disorders, trauma and stress-related disorders, etc.), or secondary depression;
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* Patients with serious or unstable diseases of the cardiovascular, liver, kidney, blood, endocrine, neurological system, and other systems or organs, especially those with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, VNS, DBS, tDCS, light therapy, or other physical therapy related to mental illness within 3 months;
* Currently receiving or planning to start formal cognitive or behavioral therapy, or systemic psychological therapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy, etc.) during the trial.
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past 1 year;
* Female of childbearing potential who plans to become pregnant during the trial.
* Female that is pregnant or breastfeeding.
* Patients in any clinical trials of other drugs or physical therapy within 1 month before the screening.
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to immediate post-treatment | Baseline, Day 5 (Immediate Post-treatment)
  The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher scores represent higher depression severity. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).

SECONDARY OUTCOMES:
Change in MADRS, HAMD-17, and QIDS_SR from baseline to different time points post-treatment | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The HAMD-17 version consists of 17 items. Higher scores represent higher depression severity. The 16-item QIDS_SR is a widely used self-report instrument covering depressive symptoms incorporating nine Diagnostic and Statistical Manual of Mental Disorder-IV (DSM-IV) diagnostic criteria for major depressive disorders. Higher scores represent higher depression severity.
Remission and response rates estimated using MADRS, HAMD, QIDS_SR | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  Three questionnaires were used to assess the response rate and remission rate of depression separately. Response is defined as an symptom improvement ≥50% on these scales; remission was defined as a score< 11 on MADRS, or <8 on HAMD, or <6 on QIDS_SR.
Safety measures using SSI and YMRS | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  Scale for Suicide Ideation (SSI) and Young Mania Rating Scale (YMRS) were used to estimated suicide ideation and manic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality, China